CLINICAL TRIAL: NCT04534309
Title: Behavioral Weight Loss for Overweight and Obese Cancer Survivors in Maryland: A Demonstration Project
Brief Title: Behavioral Weight Loss Program for Cancer Survivors in Maryland
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Maryland Cigarette Restitution Fund (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00229163
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Prostate Cancer; Melanoma (Skin); Endometrial Cancer; Gallbladder Cancer; Rectal Cancer; Kidney Cancer; Bladder Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Melanoma; Endometrial Neoplasms; Gallbladder Neoplasms; Rectal Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Directed Weight Loss with year-long weight tracking (Other): Written Weight Loss Material.
  Interventions: Behavioral: Written Weight Loss Material
- App-Directed Weight Loss with year-long weight tracking (Other): Smart phone Weight Loss App.
  Interventions: Behavioral: Weight Loss App
- Coach-Directed Weight Loss with year-long weight tracking (Other): Behavioral Lifestyle Weight Loss Intervention with Smart phone Weight Loss App.
  Interventions: Behavioral: Weight Loss App; Behavioral: Behavioral Lifestyle Weight Loss Intervention (Coaching)

INTERVENTIONS:
Behavioral: Written Weight Loss Material — Participants will receive written weight loss material by email.
  Arms: Self-Directed Weight Loss with year-long weight tracking
Behavioral: Weight Loss App — Participants will receive written weight loss material as well as instructions for using a free weight loss app on their phone or computer.
  Arms: App-Directed Weight Loss with year-long weight tracking; Coach-Directed Weight Loss with year-long weight tracking
Behavioral: Behavioral Lifestyle Weight Loss Intervention (Coaching) — Participants will receive weekly coaching phone calls to encourage regular dietary, exercise, and self-monitoring practices which encourage gradual, healthy weight loss.
  Arms: Coach-Directed Weight Loss with year-long weight tracking

SUMMARY:
Behavioral Weight Loss for Overweight and Obese Cancer Survivors in Maryland: A Demonstration Project

DETAILED DESCRIPTION:
The objective of the ASPIRE Project is to design, implement, and evaluate a real-world, lifestyle-based, support for overweight or obese cancer survivors in both urban and rural areas of Maryland. The project will provide three options of support to encourage lifestyle change to achieve and maintain a healthy weight for cancer survivors:

1. Self-Directed Weight Loss: educational materials only;
2. App-Directed Weight Loss: educational materials, weight loss app with weekly e-mail support; and
3. Coach-Directed Weight Loss: educational materials, weight loss app, weekly e-mail support and one-to-one weekly telephonic coach support.

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed with a malignant solid tumor,
* completed all required surgical, and/or chemotherapy and/or radiation curative intent therapy at least three months prior to enrollment,
* anticipated treatment-free life span of 12 months or longer.
* chemoprophylaxis with tamoxifen or aromatase inhibitors for breast cancer in women will be permitted
* anti- Luteinizing-hormone releasing therapy for prostate cancer in men will be permitted.
* BMI ≥ 25 kg/m2 (BMI ≥ 23 kg/m2 for Asians) and weight ≤ 400 lbs.
* have an email address for regular personal use

Additional criteria for participants in weight tracking (self-directed or app directed)

* willingness to record/transmit quarterly weights for 12 months

Additional criteria for App-Directed Program:

* willingness to change diet and increase physical activity and track weight, diet and physical activity
* have a smart phone for personal use
* sufficient data plan/Internet to support daily use of weight loss app*

Additional Criteria for Coach-Directed Weight Loss Program

* willingness to lose weight by changing diet and physical activity habits
* willingness to track weight, diet and physical activity
* willingness to record/transmit quarterly weights for 12 months
* smart phone for personal use
* data plan/Internet to support daily use of weight loss app*
* willingness to complete coaching calls (12 weekly calls and 3 monthly calls)
* sufficient call plan to support coaching calls

  * a corresponding website could be used, then daily Internet access is required for person use.

Exclusion Criteria:

* received any chemotherapy (unless anti-hormonal therapy) and/or radiation three months or less prior to the proposed program date
* women who are breastfeeding, pregnant, or planning pregnancy within the next year

Additional exclusion criteria for participants in weight tracking and/or Coach-Directed Program

* self-identification of uncontrolled concurrent medical condition likely to limit compliance with the program as determined by investigators.
* current involvement in another organized weight loss program
* current use of steroids or other medication known to affect body weight
* bariatric surgery scheduled within the next 6 months, or
* plan to move outside the continental US in the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Weight change at 6 months in Coach-Directed Program | Baseline and 6 months
  Evaluate the "effectiveness" of the Coach-Directed weight loss programs in a real world setting by examining weight change [in kilograms (kg)] at 6-months.

SECONDARY OUTCOMES:
Weight change at 6 months in Self-Directed and App-Directed Weight Loss Programs | Baseline and 6 months
  Evaluate the "effectiveness" of the Self-Directed and App-Directed weight loss programs in a real world setting by examining weight change [in kilograms (kg)] at 6-months.

OTHER OUTCOMES:
Program participation as assessed by participant enrollment | End of enrollment, up to 2 years
  Examine the enrollment in each program as a measure of program participation.
Adoption of weight loss program activities as assessed by app use frequency | 6 months
  Evaluate the "adoption" of the App-Directed Weight Loss Program and Coach-Directed Weight Loss Program by examining app-use frequency at six months.
Implementation of weight loss program as assessed by a participant survey | 6 months
  Evaluate the implementation of the Coach-Directed Weight Loss Program through a participant survey.
Weight change at 12 months by program | Baseline and 12 months
  Evaluate the "maintenance" of the Self-Directed, App-Directed and Coach-Directed weight loss programs in a real world setting by examining weight change [in kilograms (kg)] at 12-months by program.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Yeh, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins ProHealth, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Jerome GJ, Appel LJ, Bunyard L, Dalcin AT, Durkin N, Charleston JB, Kanarek NF, Carducci MA, Wang NY, Yeh HC. Behavioral Weight Loss Programs for Cancer Survivors Throughout Maryland: Protocol for a Pragmatic Trial and Participant Characteristics. JMIR Res Protoc. 2024 Jun 12;13:e54126. doi: 10.2196/54126. PMID 38865181